CLINICAL TRIAL: NCT02237404
Title: Sustainability of Cardiology Services: Economic Evaluation and Communication in Remote Monitoring of People With Pacemakers.
Brief Title: Economic Evaluation and Communication in Remote Monitoring of People With Pacemakers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Principal Investigator, Antonio Lopez Villegas, PhD student, University of Tromso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 008WABELCMW2014A
Record Dates: First submitted 2014-08-25; First posted 2014-09-11 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Cardiovascular Disease
Keywords: Follow-Up studies; Biological Pacemakers; Telemedicine; Efficiency
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hospital monitoring of pacemakers (No Intervention): Patients have to go to the hospital to be monitorized
- Remote monitoring of pacemakers (Experimental): Telemedicine System:
  Patients have not to go to the hospital to be monitorized
  Interventions: Device: Telemedicine System

INTERVENTIONS:
Device: Telemedicine System — Telemedicine System is used in remote monitoring group
  Other Names: Patients are monitorized from hospital
  Arms: Remote monitoring of pacemakers

SUMMARY:
The purpose of this research is to estimate the outcomes in health and cost of the follow-up of patients with pacemakers.

The initial hypothesize of this study is that remote monitoring of pacemaker will show a best relation of outcomes in costs and effectiveness than the conventional follow-up in hospital.

DETAILED DESCRIPTION:
Cardiovascular Diseases are a major cause of global morbidity and mortality, being responsible according to the World Health Organization of the 30% of overall mortality.

Since 2001 that the first pacemaker of remote monitoring was implanted in Europe, more than 300,000 pacemaker have been implanted around the world. Despite this sharp expansion, the scientific evidence on economic evaluations of pacemaker with remote monitoring is very limited, and in our knowledge, studies including informal costs have not been conducted.

In the field of cardiology, telemedicine allows consultations with patients through monitoring systems and remote communication analyzing the ongoing heart rates of people with pacemakers, implantable cardioverter defibrillators, cardiac resynchronization therapy and subcutaneous Holter. The use of remote monitoring may save time and efforts to both healthcare professionals and patients, including their informal caregivers, reducing the number of follow up visits to the hospital and reducing the associated costs with patient follow-up, which will help to improve sustainability of healthcare services.

During the 06 months of study, the patients with implant of pacemakers of both groups will be assessed of the same parameters, in 3 different moments (pre-implant and months 1, and 6 post-implantation).

Pacemakers that are going to be used in the project:

1. Remote monitoring group: Biotronik Estella SR-T and DR-T & Biotronik Evia SR-T and DR-T.
2. Hospital monitoring group: St Jude Medical Endurity SR and DR & Sorin Reply 200 SR and DR.

The study will estimate: 1) The Clinical features of the patients. 2) The effectiveness through of administration of Health-Related Quality of Life questionnaires and 3) Finally, hospital and informal costs of patients with pacemakers will be estimated by the researches.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age
* Have a pacemaker implanted
* Understand and be able to properly perform self-monitoring at home

Exclusion Criteria:

* Be participating in another study
* Refuse to participate in the study
* Have implanted a different cardiac device to the pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Clinical features | 6 months
  Selected variables from the medical history records:
  * Gender
  * Age
  * Indication for the implantation of the pacemaker.
  * Comorbidities
  * Pharmacological treatment
  * Vital signs
  * Pacemaker parameters

SECONDARY OUTCOMES:
Health-Related Quality of Life | 6 months
  EuroQol-5Dimensions (EQ-5D)
Health-Related Quality of Life | 6 months
  Minnesota Living With Heart Failure Questionnaire (MLHF)
Safety | 6 months
  * Number of patients with Adverse Events
  * Type of Adverse Events diagnosed
Consultations and Hospitalizations unscheduled | 6 months
  Number of unscheduled visits and hospitalizations
Direct costs | 6 months
  Direct costs taken into account:
  * Pacemakers' costs (device implanted)
  * Hospitalizations' costs
  * Consultations' costs (hospital)
  * Prescribed medical transport's cost
  * Health personnel costs
  * Pharmaceutical costs
Indirect cost | 6 months
  Maintenance of the medical consultation (hospital):
  * Electricity
  * Cleaning
  * Furniture
  * Health fungible
  * Equipment investment
Informal costs | 6 months
  Costs related to the care and displacements of patients to hospital:
  * Displacement costs to hospital
  * Accommodation costs
  * Cost of meals
  * Costs for caregivers

CONTACTS AND LOCATIONS:
Locations (1):
- Nordland Hospital, Bodø, Nordland, Norway

REFERENCES:
- [Derived] Lopez-Villegas A, Catalan-Matamoros D, Peiro S, Lappegard KT, Lopez-Liria R. Cost-utility analysis of telemonitoring versus conventional hospital-based follow-up of patients with pacemakers. The NORDLAND randomized clinical trial. PLoS One. 2020 Jan 29;15(1):e0226188. doi: 10.1371/journal.pone.0226188. eCollection 2020. PMID 31995558
- [Derived] Lopez-Liria R, Lopez-Villegas A, Enebakk T, Thunhaug H, Lappegard KT, Catalan-Matamoros D. Telemonitoring and Quality of Life in Patients after 12 Months Following a Pacemaker Implant: the Nordland Study, a Randomised Trial. Int J Environ Res Public Health. 2019 Jun 5;16(11):2001. doi: 10.3390/ijerph16112001. PMID 31195650
- [Derived] Lopez-Villegas A, Catalan-Matamoros D, Lopez-Liria R, Enebakk T, Thunhaug H, Lappegard KT. Health-related quality of life on tele-monitoring for users with pacemakers 6 months after implant: the NORDLAND study, a randomized trial. BMC Geriatr. 2018 Sep 21;18(1):223. doi: 10.1186/s12877-018-0911-3. PMID 30241511